CLINICAL TRIAL: NCT00040898
Title: Sho-Saiko-To After Ablation for Non-Resectable Hepatocellular Carcinoma (HCC): A Phase II Trial With Historical Control
Brief Title: Sho-Saiko-To Following Removal of Liver Cancer By Embolization in Treating Patients With Liver Cancer That Cannot Be Surgically Removed
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 01-002; P30CA008748 (NIH); MSKCC-01002; NCI-G02-2084
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Liver Cancer
Keywords: localized unresectable adult primary liver cancer; advanced adult primary liver cancer; recurrent adult primary liver cancer; adult primary hepatocellular carcinoma
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — shosaiko-to

INTERVENTIONS:
Dietary Supplement: Sho-saiko-to

SUMMARY:
RATIONALE: The Chinese herbal medicine Sho-saiko-to contains ingredients that may slow the growth of tumor cells and stimulate a person's immune system to help kill tumor cells. This may be an effective treatment following hepatic artery embolization.

PURPOSE: Phase II trial to study the effectiveness of Sho-saiko-to following hepatic artery embolization in treating patients who have liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival of patients with unresectable hepatocellular carcinoma treated with Sho-saiko-to after ablation therapy with embolization vs historical control patients.
* Compare the liver function and alpha fetoprotein levels in patients treated with this drug vs historical control patients.
* Compare the intervention-free survival in patients treated with this drug vs historical control patients.

OUTLINE: Beginning within 1 week after the first course of ablation therapy with embolization, patients receive oral Sho-saiko-to three times daily. Treatment with Sho-saiko-to continues in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 78 patients will be accrued for this study within 18-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following conditions:

  * Histologically confirmed unresectable hepatocellular carcinoma
  * Serum alpha-fetoprotein (AFP) level greater than 500 ng/mL with cirrhosis
  * Serum AFP level greater than 500 ng/mL with a liver mass and positive hepatitis B or C serology
* Receiving ablation therapy with embolization
* Extrahepatic disease allowed
* No brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 50,000/mm^3
* Hemoglobin greater than 8.0 g/dL

Hepatic:

* See Disease Characteristics
* Bilirubin less than 2.0 mg/dL
* SGOT or SGPT less than 5 times upper limit of normal (ULN)
* PT or INR less than 1.6 times ULN (if not receiving warfarin for anticoagulation)
* Albumin greater than 2.5 g/dL

Renal:

* Creatinine less than 1.8 mg/dL

Pulmonary:

* DLCO at least 50% predicted OR
* DLCO at least 70% predicted if total lung capacity less than 80% predicted
* No significant lung disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No uncontrolled infection or pain
* No other condition that would significantly impair cognitive functioning during the study
* No overt psychosis, mental disability, or other incompetency that would preclude study
* No other life-threatening illness for which the prognosis is poorer than for hepatocellular carcinoma

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent interferon

Chemotherapy:

* No prior chemotherapy within 4 weeks of initiating ablation therapy
* No concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy within 4 weeks of initiating ablation therapy
* Concurrent radiotherapy allowed

Surgery:

* See Disease Characteristics

Other:

* See Disease Characteristics
* No prior ablation therapy
* No other concurrent Sho-saiko-to or any of its constituent plants
* No other concurrent anticancer medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-01; Primary Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald DeMatteo, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States